CLINICAL TRIAL: NCT02070341
Title: A Randomized Controlled Trial Examining Patient Tolerability and Efficacy of Bowel Preparation With Split Dose Picosalax vs. Split Dose Polyethylene Glycol
Brief Title: Patient Tolerability and Efficacy of Bowel Preparation With Split Dose Picosalax vs. Split Dose PEG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant changes to protocol and study design, study stopped to further enrollment and new study designed.
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Hookey Picosalax PEG
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Bowel Preparation
Keywords: patient tolerability; quality
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Split dose PEG (Experimental): Patients randomized to the Polyethylene Glycol (PEG) group will be instructed to ingest 2L of bowel preparation the night before their colonoscopy (starting at 7PM), as well as 1.5-2L of carbohydrate-electrolyte rehydration solution. The following day they will be instructed to ingest the remaining 2L of bowel preparation and must finish ingesting the entire preparation at least 4 hours prior to the scheduled colonoscopy.
  Interventions: Drug: Polyethylene Glycol
- Split dose Picosalax (Experimental): Patients randomized to the Picosalax (P/MC) group will be instructed to mix one sachet in 150mL of water and ingest the entire mixture at 7PM the night before their colonoscopy. In addition, they will be instructed to ingest 1.5-2L of carbohydrate-electrolyte rehydration solution after they consume the P/MC sachet. The following day they will mix the second sachet in 150mL of water and must finish ingesting the entire preparation at least 4 hours prior to the scheduled colonoscopy. They will also be instructed to drink additional carbohydrate-electrolyte rehydration solution after they ingest the P/MC sachet.
  Interventions: Drug: Picosalax

INTERVENTIONS:
Drug: Polyethylene Glycol
  Arms: Split dose PEG
Drug: Picosalax
  Arms: Split dose Picosalax

SUMMARY:
Introduction: Colonoscopy is an important tool for colon cancer screening. Proper colon cleansing is essential to ensure adequate mucosal examination. Timing of bowel preparation administration is now recognized as an important component for achieving superior cleansing. Multiple randomized controlled trials and meta-analyses have found split-dosing to be superior than day-before dosing. Objective: This study aims to compare two types of bowel preparations in split-doses to assess for differences in patient tolerability, as well as efficacy of colon cleansing. Methods: This is a prospective, single-blinded, randomized-controlled trial. Patients who are being referred for a colonoscopy will be recruited to participate in the study. They will be randomly assigned to receive either a split-dose polyethylene glycol (PEG) or picosalax (P/MC) bowel preparation. Patient tolerability will be examined through questionnaires. The endoscopist performing the colonoscopy will use two standardized bowel preparation scoring systems to evaluate the quality of the cleansing. The investigators propose that P/MC will be superior to PEG in patient tolerability and non-inferior in bowel cleansing effects.

ELIGIBILITY:
Inclusion Criteria:

* All male and non-pregnant female patients between ages 18 and 75 years old who require outpatient colonoscopy

Exclusion Criteria:

* ileus or bowel obstruction, previous colorectal surgery, ascites, recognized renal impairment, defined as GFR less than normal in 3 months prior to enrollment, active inflammatory bowel disease, insulin dependent diabetes, pregnancy, or recent (<6 months) myocardial infarction or unstable angina

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Patient tolerability | Two days
  Patients will be asked to complete a questionnaire to assess ease of completion and symptoms. Questionnaire items are weighted on a 5-point Likert scale. Interference with sleep will be assessed through a questionnaire that is based on a modified validated sleep questionnaire (St. Mary's Hospital Sleep Questionnaire). Participants will be asked to complete this questionnaire at the initial appointment and again on the day of their procedure

SECONDARY OUTCOMES:
Quality of bowel preparation | During colonoscopy
  The colonoscopist will be blinded to the type of preparation the subject underwent. The colonoscopist will complete a validated questionnaire to assess the quality of the preparation (The Ottawa Scale) and the 4-point Aronchick bowel cleansing scale. The patient's baseline bowel habit will be recorded, as well as the withdrawal time, volume of liquid suctioned and volume of washing fluid used during the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, Principal Investigator — Queen's University; Stephen Vanner, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada